CLINICAL TRIAL: NCT00741000
Title: The Effects of Cervical Stairstep on Cervical Range of Motion
Brief Title: Cervical Stairstep and Effects on Range of Motion (ROM)
Acronym: CSEROM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Mary Unger-Boyd, DC, Logan College of Chiropractic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SR0331080127
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Range of Motion, Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Cervical low force mobilization procedure.
  Interventions: Procedure: Cervical Stairstep

INTERVENTIONS:
Procedure: Cervical Stairstep — Cervical low force mobilization procedure.

SUMMARY:
Observe the effects of Cervical Stairstep on Cervical Spine Range of Motion

DETAILED DESCRIPTION:
The cervical spine can be affected in a number of ways due to its vulnerability to injury. These injuries can result from poor posture, sports or occupation and can lead to degenerative changes. Cervical range of motion (ROM) is also affected by these injuries. When active ROM is restricted, the injury is of muscular origin. Pain with passive ROM indicates ligamentous injury whereas restricted passive ROM indicates blockage within bone or soft tissue. The normal range of motion in the cervical spine is 80-90 degrees flexion, 70 degrees extension, 20-45 degrees lateral flexion and 90 degrees of rotation. A common mechanism of cervical spine injury is axial loading. Axial loading can create a buckling effect within the cervical spine and decrease its ability to move normally, creating a limited ROM.

ELIGIBILITY:
Inclusion Criteria:

* students and faculty between ages 18 and 50

Exclusion Criteria:

* current neck pain (as measured by the Neck Disability Index (NDI) and utilizing Jackson's and maximal foraminal compression tests to assess for radiating symptoms)
* severe recent head trauma
* acute exacerbations within the past 3 months
* known cervical disc problems
* surgical fusions within the cervical spine
* highly acute symptoms
* a positive valsalva test
* seizure disorder
* analgesics
* muscle relaxants
* medications with effects on the musculoskeletal system
* chiropractic manipulation within 48 hours of the study
* Other exclusions can be made based on investigator judgment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Cervical Range of Motion | Pre and post treatment

SECONDARY OUTCOMES:
Neck Disability Index | pre and post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Logan University, College of Chiropractic, Chesterfield, Missouri, United States